CLINICAL TRIAL: NCT04314895
Title: Phase 2 Trial Evaluating the Safety and Tolerability of Intratumoral Injections of NanoPac® With Standard of Care Therapy in Subjects With Lung Cancer
Brief Title: Trial of NanoPac Intratumoral Injection in Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NanOlogy, LLC (Industry)
Collaborators: US Biotest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NANOPAC-2020-01
Expanded Access: NCT03756311 (No longer available)
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer, Nonsmall Cell; Lung Cancer; Lung Cancer, Small Cell; Neoplasm of Lung
Keywords: paclitaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Powders; Suspensions; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NanoPac (Experimental): Intratumoral injection of NanoPac 15 mg/mL at a volume of up to 20% of the total calculated tumor and lymph node volume (not to exceed 40 mL) on up to three occasions 4 weeks apart.
  Interventions: Drug: NanoPac (sterile nanoparticulate paclitaxel) Powder for Suspension

INTERVENTIONS:
Drug: NanoPac (sterile nanoparticulate paclitaxel) Powder for Suspension — NanoPac is manufactured using a Precipitation with Compressed Antisolvent (PCA) technique that employs supercritical carbon dioxide and acetone to generate paclitaxel nanoparticles within a well-characterized particle-size distribution. Following PCA, NanoPac is filled into a clear 60mL Type 1, USP, clear-glass vial (306 mg/vial) as a powder fill of nanoparticulate paclitaxel, closed with a bromobutyl rubber stopper and aluminum crimp seal, and sterilized by gamma irradiation. Prior to administration at the hospital/clinic, NanoPac will be reconstituted with 1% Polysorbate 80, NF in 0.9% Sodium Chloride for Injection, USP, to form a suspension. The suspension will be further diluted with 0.9% Sodium Chloride for Injection, USP to achieve the final clinical formulation.
  Other Names: paclitaxel

SUMMARY:
This study evaluates the use of NanoPac injected directly into tumors in the lung of people with lung cancer.

DETAILED DESCRIPTION:
NanoPac is very small (submicron) particles of the chemotherapy drug, paclitaxel, which is administered intravenously in a number of types of cancer. These submicron particles are injected directly into solid tumors to target cancer at the site of disease with less systemic exposure than intravenously administered chemotherapy. In this study, the submicron particle paclitaxel will be injected directly into tumors in the lungs of people with small cell or non-small cell lung cancer. All subjects in this study will receive NanoPac and will be evaluated to see if NanoPac is safe and has an effect on the tumor within the lung.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Age ≥18 years and able to tolerate the EBUS-TBNI procedure;
* Histologically/cytologically confirmed lung cancer. Eligible subjects may include, for example: primary or recurrent non-resectable disease, locally advanced stages II and III with nodal disease, stage IV advanced disease;
* At least one lesion documented via imaging (within 4 weeks of Screening) which can be accessed using EBUS-TBNI;
* Subject is not a candidate for surgery;
* Has received or plans to receive SOC chemotherapy; adequate hematologic recovery must be confirmed according to the institution's SOC;
* Performance Status (ECOG) 0-2 at study entry;
* Life expectancy of at least 6 months;
* Adequate marrow, liver, and renal function at study entry;

  * ANC ≥ 1.5 x 109/L;
  * Hemoglobin ≥ 9.0 grams/dL;
  * Platelets ≥ 75 x 109/L;
  * Total bilirubin ≤ 1.5x institutional ULN;
  * AST/ ALT ≤ 2.5x institutional ULN;
  * Creatinine ≤ 1.5x institutional ULN;
* Appropriate steps taken to minimize or avoid the potential for pregnancy for subjects of child-bearing potential.*

Exclusion Criteria:

* Significant cardiac disease (Class III or IV per New York Heart Association guidelines);
* Active bacterial, viral, or fungal infections (including active AIDS, hepatitis B or hepatitis C);
* Symptomatic central nervous system (CNS) metastasis which are neurologically unstable, or CNS disease requiring increase in steroid dose (treated metastatic disease and stable steroid use are not excluded)
* Known hypersensitivity to study agent;
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shelagh Verco, PhD, Study Director — US Biotest, Inc.
Locations (4):
- United States (4):
  - University of Florida Health, Gainesville, Florida
  - Parkview Research Institute, Fort Wayne, Indiana
  - Johns Hopkins, Baltimore, Maryland
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NanoPac 15 mg/mL: Intratumoral injection of NanoPac 15 mg/mL at a volume of up to 20% of the total calculated tumor and lymph node volume (not to exceed 40 mL) on up to three occasions 4 weeks apart.
Period: Overall Study
Arm/Group | NanoPac 15 mg/mL
Started | 18
One Injection | 3
Two Injections | 5
Three Injections | 10
Completed | 5
Not Completed | 13
Not completed — Lost to Follow-up | 1
Not completed — Death | 10
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | NanoPac 15 mg/mL
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 68.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Type of Lung Cancer [Count of Participants; unit: Participants]
  Adenocarcinoma | 8
  Squamous cell carcinoma | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: AEs were collected at all study visits from the time of dosing. Subjects were required to spontaneously report any AE. Study personnel asked open-ended questions to obtain information about AEs at every visit.
Time Frame: Day 1 to Week 24 (6 Months)
Population: All subjects enrolled provided data for this outcome measure.
  Of the 18 subjects enrolled, one subject in the "NanoPac 15 mg/ml - One Injection" arm was determined to have non-malignant disease after pathology review following initial injection with NanoPac, and this subject is therefore not included in efficacy assessments but was included in the outcome measure of number of participants with treatment emergent adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | NanoPac 15 mg/mL
Number analyzed (Participants) | 18
Participants | 18

2. Secondary Outcome: Concentration of Paclitaxel in the Systemic Circulation Post-injection
Description: To characterize the pharmacokinetics of intratumoral NanoPac, plasma samples were taken on days of NanoPac injection prior to injection and at 1, 2, and 4 hours after NanoPac injection, as well as at all other study visits up through Week 24. Plasma paclitaxel concentrations are reported in pg/mL.
Time Frame: Day 1, Weeks 1, 2, 4, 5, 6, 8, 9, 10, 12, 18, and 24
Population: Of the 18 subjects enrolled, one subject in the "NanoPac 15 mg/ml - One Injection" arm was determined to have non-malignant disease after pathology review following initial injection with NanoPac, and this subject is therefore not included in efficacy assessments but was included in the outcome measure of concentration of paclitaxel in the systemic circulation post-injection. The remaining two subjects in the "NanoPac 15 mg/ml - One Injection" arm discontinued from the study prior to Week 12.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- NanoPac 15 mg/mL - One Injection: Intratumoral injection of NanoPac 15 mg/mL at a volume of up to 20% of the total calculated tumor and lymph node volume (not to exceed 40 mL) on up to three occasions 4 weeks apart. These subjects received only one of the optional three NanoPac injections.
- NanoPac 15 mg/mL - Two Injections: Intratumoral injection of NanoPac 15 mg/mL at a volume of up to 20% of the total calculated tumor and lymph node volume (not to exceed 40 mL) on up to three occasions 4 weeks apart. These subjects received two of the optional three NanoPac injections.
- NanoPac 15 mg/mL - Three Injections: Intratumoral injection of NanoPac 15 mg/mL at a volume of up to 20% of the total calculated tumor and lymph node volume (not to exceed 40 mL) on up to three occasions 4 weeks apart. These subjects received all three of the optional NanoPac injections.
Arm/Group | NanoPac 15 mg/mL - One Injection | NanoPac 15 mg/mL - Two Injections | NanoPac 15 mg/mL - Three Injections
Number analyzed (Participants) | 3 | 5 | 10
pg/mL
  Day 1 - Pre-Injection | 566.7 (981.50) | 44.2 (82.61) | 32.8 (103.72)
  Day 1 - 1 Hr Post-Injection: number analyzed (Participants) | 2 | 5 | 10
  Day 1 - 1 Hr Post-Injection | 10685.0 (3415.33) | 24104.0 (28642.55) | 45523.7 (93639.03)
  Day 1 - 2 Hr Post-Injection: number analyzed (Participants) | 2 | 5 | 10
  Day 1 - 2 Hr Post-Injection | 6470.0 (2757.72) | 21850.0 (20982.28) | 27678.1 (49332.88)
  Day 1 - 4 Hr Post-Injection: number analyzed (Participants) | 2 | 4 | 9
  Day 1 - 4 Hr Post-Injection | 4360.0 (1767.77) | 9877.5 (8798.58) | 25884.8 (46389.73)
  Week 1: number analyzed (Participants) | 1 | 4 | 10
  Week 1 | 2070.0 (NA) — Only 1 subject provided plasma in this group at this timepoint | 3232.0 (2284.86) | 2399.3 (3981.41)
  Week 2: number analyzed (Participants) | 2 | 5 | 9
  Week 2 | 810.0 (1145.51) | 1739.0 (2011.08) | 10215.3 (28268.21)
  Week 4 - Pre-Injection: number analyzed (Participants) | 1 | 4 | 10
  Week 4 - Pre-Injection | 0.0 (NA) — Only 1 subject provided plasma in this group at this timepoint | 2125.3 (2056.14) | 863.7 (1319.34)
  Week 5: number analyzed (Participants) | 0 | 3 | 8
  Week 5 |  | 2662.0 (1977.22) | 1933.5 (3036.68)
  Week 6: number analyzed (Participants) | 1 | 2 | 9
  Week 6 | 1060.0 (NA) — Only 1 subject provided plasma in this group at this timepoint | 21640.0 (28369.12) | 1357.1 (2031.87)
  Week 8 - Pre-Injection: number analyzed (Participants) | 1 | 3 | 10
  Week 8 - Pre-Injection | 0.0 (NA) — Only 1 subject provided plasma in this group at this timepoint | 7976.3 (12147.98) | 702.5 (1171.64)
  Week 9: number analyzed (Participants) | 0 | 2 | 8
  Week 9 |  | 17695.0 (16977.63) | 1951.5 (4991.29)
  Week 10: number analyzed (Participants) | 0 | 1 | 7
  Week 10 |  | 11900.0 (NA) — Only 1 subject provided plasma in this group at this timepoint | 1813.1 (2291.70)
  Week 12: number analyzed (Participants) | 1 | 2 | 8
  Week 12 | 667.0 (NA) — Only 1 subject provided plasma in this group at this timepoint | 7953.5 (10955.21) | 551.9 (980.98)
  Week 18: number analyzed (Participants) | 1 | 2 | 6
  Week 18 | 0.0 (NA) — Only 1 subject provided plasma in this group at this timepoint | 4910.5 (6801.66) | 80.7 (176.92)
  Week 24: number analyzed (Participants) | 1 | 2 | 5
  Week 24 | 589.0 (NA) — Only 1 subject provided plasma in this group at this timepoint | 5770.1 (8103.37) | 10.6 (23.75)

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) as assessed using RECIST v1.1
Time Frame: Weeks 24, 38, and 52
Population: Of the 18 subjects enrolled, one subject was determined to have non-malignant disease after pathology review following initial injection with NanoPac, and this subject is therefore not included in efficacy assessments i.e. PFS.
Measure: Count of Participants; unit: Participants
Arm/Group | NanoPac 15 mg/mL - One Injection | NanoPac 15 mg/mL - Two Injections | NanoPac 15 mg/mL - Three Injections
Number analyzed (Participants) | 2 | 5 | 10
Participants
  Week 24: Progression Free | 0 | 0 | 5
  Week 24: Progressed or Died | 2 | 5 | 4
  Week 24: Censored | 0 | 0 | 1
  Week 38: Progression Free | 0 | 0 | 4
  Week 38: Progressed or Died | 2 | 5 | 5
  Week 38: Censored | 0 | 0 | 1
  Week 52: Progression Free | 0 | 0 | 2
  Week 52: Progressed or Died | 2 | 5 | 6
  Week 52: Censored | 0 | 0 | 2

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) as determined by survival time following first NanoPac injection
Time Frame: Weeks 24, 38, and 52
Population: Of the 18 subjects enrolled, one subject was determined to have non-malignant disease after pathology review following initial injection with NanoPac, and this subject is therefore not included in efficacy assessments i.e. overall survival.
Measure: Count of Participants; unit: Participants
Arm/Group | NanoPac 15 mg/mL - One Injection | NanoPac 15 mg/mL - Two Injections | NanoPac 15 mg/mL - Three Injections
Number analyzed (Participants) | 2 | 5 | 10
Participants
  Week 24: Confirmed Alive | 0 | 3 | 6
  Week 24: Dead | 1 | 2 | 3
  Week 24: Censored | 1 | 0 | 1
  Week 38: Confirmed Alive | 0 | 3 | 4
  Week 38: Dead | 1 | 2 | 5
  Week 38: Censored | 1 | 0 | 1
  Week 52: Confirmed Alive | 0 | 1 | 2
  Week 52: Dead | 1 | 3 | 6
  Week 52: Censored | 1 | 1 | 2

5. Secondary Outcome: Change in Tumor Dimensions (Longest Diameter)
Description: Change in longest dimension (cm) as determined by CT imaging compared to baseline (Screening)
Time Frame: Weeks 12, 24, 38, and 52
Population: Of the 18 subjects enrolled, one subject in the "NanoPac 15 mg/ml - One Injection" arm was determined to have non-malignant disease after pathology review following initial injection with NanoPac, and this subject is therefore not included in efficacy assessments, i.e. change in tumor dimensions (longest diameter). The remaining two subjects in the "NanoPac 15 mg/ml - One Injection" arm discontinued from the study prior to Week 12.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | NanoPac 15 mg/mL - One Injection | NanoPac 15 mg/mL - Two Injections | NanoPac 15 mg/mL - Three Injections
Number analyzed (Participants) | 0 | 5 | 10
cm
  Week 12 - Change from Baseline: number analyzed (Participants) | 0 | 2 | 6
  Week 12 - Change from Baseline |  | 2.06 (2.913) | -0.23 (0.907)
  Week 24 - Change from Baseline: number analyzed (Participants) | 0 | 2 | 6
  Week 24 - Change from Baseline |  | 1.26 (1.216) | -0.78 (0.678)
  Week 38 - Change from Baseline: number analyzed (Participants) | 0 | 1 | 4
  Week 38 - Change from Baseline |  | 1.0 (NA) — Data available from only one subject | -0.85 (0.635)
  Week 52 - Change from Baseline: number analyzed (Participants) | 0 | 1 | 3
  Week 52 - Change from Baseline |  | 1.62 (NA) — Data available from only one subject | -0.91 (0.753)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was assessed through study completion, up to 52 weeks; all adverse events were collected from the time of dosing until Week 24.
Description: AEs were collected at all study visits from the time of dosing. Subjects were required to spontaneously report any AE. Study personnel asked open-ended questions to obtain information about AEs at every visit.
Arm/Group | NanoPac 15 mg/mL - One Injection | NanoPac 15 mg/mL - Two Injections | NanoPac 15 mg/mL - Three Injections
All-Cause Mortality (participants affected / at risk) | 1/3 | 3/5 | 6/10
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/5 | 7/10
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NanoPac 15 mg/mL - One Injection (N=3) | NanoPac 15 mg/mL - Two Injections (N=5) | NanoPac 15 mg/mL - Three Injections (N=10)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Fluid overload (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NanoPac 15 mg/mL - One Injection (N=3) | NanoPac 15 mg/mL - Two Injections (N=5) | NanoPac 15 mg/mL - Three Injections (N=10)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Adrenal mass (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (7)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 5 (5)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (3) | 0 (0) | 2 (3)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (2)
Fatigue (General disorders) | 2 (2) | 3 (3) | 4 (4)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 5 (6)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Systemic candida (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural oedema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Clubbing (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changed (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT04314895/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/95/NCT04314895/SAP_001.pdf